CLINICAL TRIAL: NCT07232056
Title: Geriatric Oncology Assessment to Link With Support for Older Women Taking Adjuvant Aromatase Inhibitor Therapy
Brief Title: Geriatric Oncology Assessment and Coping Skills Training for Older Women on Aromatase Inhibitor Therapy
Acronym: GOAL-AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00118528
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer, Hormone Receptor Positive, Aromatase Inhibitor-Associated Arthralgia
Keywords: Breast Neoplasms; Geriatric Oncology; Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GOAL-AI + CST-AI (Experimental): Combination of clinic-level geriatric assessment and CBT-based coping skills training.
  Interventions: Behavioral: GOAL-AI; Behavioral: CST-AI
- GOAL-AI alone (Experimental): Clinic-level geriatric assessment and support only.
  Interventions: Behavioral: GOAL-AI
- CST-AI alone (Experimental): CBT-based coping skills training only.
  Interventions: Behavioral: CST-AI
- Enhanced Usual Care (No Intervention): Standard care with educational materials.

INTERVENTIONS:
Behavioral: GOAL-AI — Clinic-level geriatric assessment and support program.
  Arms: GOAL-AI + CST-AI; GOAL-AI alone
Behavioral: CST-AI — CBT-based coping skills training via telehealth.
  Arms: CST-AI alone; GOAL-AI + CST-AI

SUMMARY:
Older women (≥65 years) with HR+ non-metastatic breast cancer experience high symptom burden and reduced quality of life during aromatase inhibitor (AI) therapy. This hierarchical 2×2 factorial randomized controlled trial will test two interventions: (1) a clinic-level geriatric oncology assessment and support program (GOAL-AI) and (2) a patient-level CBT-based coping skills training (CST-AI). The study aims to improve pain, symptom burden, and health-related quality of life compared to enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* Female, age ≥65 years
* HR+ non-metastatic breast cancer
* Within 12 months of starting AI therapy
* English-speaking
* Able to provide consent

Exclusion Criteria:

* Age <65 years
* Metastatic cancer
* Cognitive impairment preventing consent
* Receiving care at multiple participating sites

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity and interference as measured by the Brief Pain Inventory - Short Form | Baseline, 6 months, 12 months
  The Brief Pain Inventory-Short Form (BPI-SF) will be used to assess pain severity and interference from pain across important life domains (e.g., general activity, work, relations with others). To calculate a pain severity score, the BPI-SF averages worst, least, average and current pain severity ratings on a 0 to 10 scale, with higher scores indicating more severe pain. To calculate a pain interference score, 7 items asking about interference from pain across different life domains will be averaged, with higher scores indicating higher pain interference.

SECONDARY OUTCOMES:
Change in emotional distress, as measured by the PROMIS® Anxiety and Depression 4-item Short Forms | Baseline, 6 months, 12 months
  For the PROMIS® Anxiety and Depression 4-item Short Forms (4a, v1.0) items are summed to create a raw score from 4 to 20 that is converted to a T-score. Responses are on a 5-point scale from "never" (1) to "always" (5). Higher scores indicate higher emotional distress.
Change in fatigue, as measured by the PROMIS® Fatigue 6-item Short Form | Baseline, 6 months, 12 months
  For the PROMIS® Fatigue 6-item Short Form (6a, v1.0) items are summed to create a raw score that is converted to a T-score. Participants are asked to think about the last week when responding to each item (e.g., "In the past 7 days, how run-down did you feel, on average?"), providing ratings on a scale from "not at all" (1) to "very much" (5). Sum scores may range from 6 to 30, with higher scores indicating higher fatigue.
Change in physical function, as measured by the Five Times Sit to Stand Test (5xSST) | Baseline, 6 months, 12 months
  The Five Times Sit to Stand Test (5xSST) assesses functional lower extremity strength, balance, risk of fall, functional decline, and frailty. The amount of time it takes a patient to sit and stand five times in succession with arms folded across their chest is averaged across three trials.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shelby, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: Yes
The following data will be preserved and shared: patient-reported data from study assessments, healthcare utilization data collected from the health record, AI adherence data collected via self-report and from the health record, physical function and geriatric assessment data collected by study staff in clinic and from the health record, and socio-demographic and medical data collected via patient report and health record.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared either at the time of publication or at the end of the performance period, whichever comes first. All data deposited with the Duke Research Data Repository will be retained for a minimum of 25 years according to their stated Retention Policy.